CLINICAL TRIAL: NCT04364750
Title: Biomarkers of Diet-microbiota Interactions in Irritable Bowel Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: BFIBS
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: FODMAP; microbiota; histamine
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Histidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Participants in group A will undergo challenges in the order:
  1. High-FODMAP beverage + placebo probiotic + L-Histidine
  2. Low-FODMAP beverage + placebo probiotic + L-Histidine
  3. High-FODMAP beverage + probiotic + L-Histidine
  Challenges each last 5 days, but the FODMAP drinks and the L-Histidine capsules are only taken for the last three days. There is a 10 day washout period between challenges.
  Interventions: Dietary Supplement: L-Histidine; Dietary Supplement: High-FODMAP beverage; Dietary Supplement: Low-FODMAP beverage; Dietary Supplement: Lactobacillus acidophilus CL1285, L. casei LBC80R and L. rhamnosus CLR2.; Other: Placebo
- Group B (Experimental): Participants in group A will undergo challenges in the order:
  1. Low-FODMAP beverage + placebo probiotic + L-Histidine
  2. High-FODMAP beverage + probiotic + L-Histidine
  3. High-FODMAP beverage + placebo probiotic + L-Histidine.
  Challenges each last 5 days, but the FODMAP drinks and the L-Histidine capsules are only taken for the last three days. There is a 10 day washout period between challenges.
  Interventions: Dietary Supplement: L-Histidine; Dietary Supplement: High-FODMAP beverage; Dietary Supplement: Low-FODMAP beverage; Dietary Supplement: Lactobacillus acidophilus CL1285, L. casei LBC80R and L. rhamnosus CLR2.; Other: Placebo
- Group C (Experimental): Participants in group A will undergo challenges in the order:
  1. High-FODMAP beverage + probiotic + L-Histidine
  2. High-FODMAP beverage + placebo probiotic + L-Histidine
  3. Low-FODMAP beverage + placebo probiotic + L-Histidine.
  Challenges each last 5 days, but the FODMAP drinks and the L-Histidine capsules are only taken for the last three days. There is a 10 day washout period between challenges.
  Interventions: Dietary Supplement: L-Histidine; Dietary Supplement: High-FODMAP beverage; Dietary Supplement: Low-FODMAP beverage; Dietary Supplement: Lactobacillus acidophilus CL1285, L. casei LBC80R and L. rhamnosus CLR2.; Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-Histidine — 1 capsule (0.6g) twice daily
Dietary Supplement: High-FODMAP beverage — High-FODMAP beverage (10g of fermentable carbohydrates) consumed twice daily.
Dietary Supplement: Low-FODMAP beverage — Low-FODMAP beverage (10g glucose) consumed twice daily.
Dietary Supplement: Lactobacillus acidophilus CL1285, L. casei LBC80R and L. rhamnosus CLR2. — Total of 50 billion CFU/capsule taken twice daily.
  Other Names: Bio-K+ 50 Billion
Other: Placebo — Enteric coated capsule with no active ingredient, taken twice daily

SUMMARY:
Most patients suffering from the irritable bowel syndrome (IBS) report that ingestion of certain foods is a major trigger of symptoms, but the reason is unclear. Previous studies have shown that foods containing poorly absorbed carbohydrates (FODMAPs) are fermented by the bacteria in our bowels and these cause symptoms in some but not all patients. Gut bacteria are capable of producing various products, such as neuroimmune mediator histamine, that may be related to IBS symptoms. Our recent data suggest that consumption of FODMAPs promotes production of bacterial histamine.

The main objective of this study is to investigate bacterial production of histamine and its relationship to IBS symptoms. The study will involve 6 weeks on a low-FODMAP diet with three three-day interventions consisting of High- or Low-FODMAP drinks along with probiotics or placebo capsules. The patient's bacteria and metabolites will be analyzed at various time points.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 with IBS (Rome IV criteria) who have self-reported previous improvement in their IBS symptoms while on a low FODMAP diet, or when excluding certain high-FODMAP foods, or patients in whom histamine is expected to play a key role (either diagnosed with high histamine producing bacteria, or improved IBS symptoms after using antihistamines). Individuals should be able to swallow size 00 capsules.

Exclusion Criteria:

* Concurrent significant organic GI pathology (i.e. celiac, IBD, etc.)
* Concurrent systemic disease (such as diabetes) and/or laboratory abnormalities considered by investigators to be risky or that could interfere with data collection
* History of active cancer in the last 5 years, other than basal cell cancer
* Pregnant or breastfeeding women
* Active or recent participation (< 1 month) in a clinical study, except for SPOR IMAGINE
* Use of antibiotics, probiotics, or ACE inhibitors during, or one month prior to the study
* Use of new medications less than 4 weeks prior to the study.
* Allergies to any of the ingredients used in the study
* Any immune-compromising conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Metabolites in stool, urine and blood | six weeks
  Metabolites will be measured by LC-MS and ELISA at baseline and before and after each intervention.

SECONDARY OUTCOMES:
Expression of hdc gene by stool bacteria | six weeks
  Gram-positive and Gram-negative bacteria will be assessed by PCR using custom designed primers
Stool microbiota composition | six weeks
  16S rRNA Illumina sequencing of stool samples with culture-enriched sequencing.
Worsening of IBS symptoms following High-FODMAP challenge | six weeks
  Increase by ≥50 points on IBS Symptom Severity Score (IBS-SSS). The score will be used as a dichotomous variable. The overall score ranges from 0 to 500, with higher scores indicating greater symptom severity.
Changes in IBS symptoms | six weeks
  IBS-SSS continuous data. The overall score ranges from 0 to 500, with higher scores indicating greater symptom severity.
Changes in general GI symptoms | six weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) for general GI symptoms. Four subscales will be used: Gas & Bloating, Diarrhea, Constipation, and Belly Pain. T-scores are calculated using the Scoring Service by Health Measures and range from 34.7 - 79.0 (Gas & Bloating), 39.9 - 75.2 (Diarrhea), 40.6 - 80.8 (Constipation), and 33.9 - 80.0 (Belly Pain). On this scale, 50 indicates the mean of the general population and a difference of 10 is a standard deviation. Higher scores indicate greater symptom severity.
Levels of anxiety, depression and stress | six weeks
  Depression Anxiety Stress Scale (DASS-21) to assess psychiatric comorbidity and stress. The scale scores range from 0 - 42 with higher scores indicating worse outcomes.
Changes in dietary intake | six weeks
  5-day food diaries will be completed at 5 time points. FODMAP intake will be quantified using Monash University software and database

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Bercik, MD, Principal Investigator — McMaster University; Stephen Vanner, MD, Principal Investigator — Queens University
Locations (2):
- Canada (2):
  - McMaster University Medical Centre, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No